CLINICAL TRIAL: NCT00421226
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Demonstrate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ACZ885 Administered as Intravenous Infusion and Subcutaneous Injection in Japanese Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ACZ885 in Healthy Japanese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885A1101
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Safety, tolerability, pharmacokinetics, pharmacodynamics, ACZ885, Japanese,
MeSH Terms: interventions — canakinumab

INTERVENTIONS:
Drug: ACZ885

SUMMARY:
This study will evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of ACZ885 administered via intravenous infusion and subcutaneous injection in healthy Japanese male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy male subjects age 20 to 45 years of age, and in good health
* At screening and baseline, the subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis.
* Body mass index within the range of 18 to 28 kg/m2 and weigh 50 to 100 kg

Exclusion Criteria:

* Smokers.
* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing. Acetaminophen is acceptable. Treatment of any biologics within three months prior to dosing. Having live vaccinations within six months prior to dosing.
* Participation in any clinical investigation within 4 months prior to dosing.
* Donation or loss of 400 mL or more of blood within 3 months; donation or loss of 200 mL or more of blood within 1 month; or donation of component blood within 2 weeks prior to participation.
* Significant illness (sinusitis, pneumonia, cystitis, sepsis, etc) within two weeks prior to dosing.
* A past personal or close family medical history of cardiac disorders
* History of:

  * fainting,
  * low blood pressure when standing,
  * abnormal heart rhythms
  * acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* Clinically significant drug allergy or history and complication of atopic allergy (asthma, urticaria, eczematous dermatitis)
* Known hypersensitivity to the study drug or similar drugs
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or jeopardize participation in the study.
* History of immunodeficiency diseases, including a positive HIV test result.
* A positive Hepatitis B surface antigen (HBsAg), Hepatitis C or Syphilis test result.
* Drug or alcohol abuse within the 12 months prior to dosing
* Tuberculosis symptoms, complication of tuberculosis, contact with patients with suspected tuberculosis symptoms

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative site, Tokyo, Japan